CLINICAL TRIAL: NCT05748951
Title: A Pilot Clinical Evaluation of Canalicular Occlusion
Brief Title: Evaluating a Device for Blocking the Tear Duct
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: AesculaTech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TP-0183-01
Record Dates: First submitted 2023-02-18; First posted 2023-03-01 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tear Duct Plug (Experimental): A device inserted into the tear duct to block tear drainage
  Interventions: Device: Canalicular occlusion device

INTERVENTIONS:
Device: Canalicular occlusion device — Occlusive device is inserted into the tear duct to block tear drainage

SUMMARY:
Participants will receive a tear duct plug to see if their eye comfort improves.

DETAILED DESCRIPTION:
Participants will receive a canalicular occlusion and will be followed for 3 months so that safety and effectiveness of the device may be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 22 or older complaining of ocular dryness who report having to use artificial tears or lubricants.
2. Both of the following conditions:

   * Baseline symptoms score of 23 or higher on the OSDI questionnaire; and
   * OSDI Questionnaire has 3 or fewer responses of "not applicable"
3. Basal tear secretion (Schirmer I Test with anesthesia) < 10mm/5 minutes (in one of the two eyes). The eye with the lower score is the study eye.
4. Willing and able to comply with the study procedures and follow-up.
5. Willing and able to provide informed consent.

Exclusion Criteria:

1. Presence or history of chronic or current, acute ocular inflammation or infection, aside from mild blepharitis or inflammation associated with primary dry eye or disorders which are known to cause dry eyes (e.g. Sjrögens Syndrome).
2. The presence of any lacrimal occlusion, ocular disorder, or condition in either eye, conjunctiva, or lacrimal system that, in the opinion of the investigator, would interfere with the interpretation of the study results (e.g., corneal transplant, routine ocular injections, recent ocular surgery, ectropion, surgical procedure such as cautery, or past canalicular surgery, significant corneal or conjunctival scarring, pterygium or nodular pinguecula; active ocular herpetic infection; lid or lacrimal cancer; clinically significant corneal dystrophy or other disorder which may cause rapid degeneration of visual acuity, such as anterior (epithelial) basement membrane corneal dystrophy, clinical keratoconus, or active, wet macular degeneration.
3. Presence of - or unverified removal of - other canalicular occlusion devices.
4. Chronic allergic rhinitis
5. Allergic to study materials, supplies and medication.
6. Contraindication to topical anesthesia.
7. Actively using a topical medication (such as steroids and immunosuppressants) for which the use of a plug may cause complications, regardless of dosage adjustment.
8. Participation in another ophthalmic clinical trial within three months prior to enrollment. Participant must also be willing to refrain from another ophthalmic study for the duration of the study.
9. Co-existing health condition(s), either ocular or non-ocular that, in the judgement of the investigator could affect the safety or effectiveness of treatment, the compliance of the participant to the protocol, or other factors which may confound validity of study data collection or analysis. For example, participants who are pregnant or nursing, have pterygium, or uncontrolled blepharitis for which artificial lubricants do not provide relief are excluded. Unless post-menopausal or medically sterile (e.g hysterectomy, bilateral tubal ligation, bilateral oophorectomy), female participants must have a negative urine pregnancy test (UPT) on Day 0 of the study and should utilize a medically acceptable form of contraception over the course of the study.
10. Use of drugs under any of the following conditions:

    * Change in dry eye medication (e.g., Restasis or Xiidra) within 60 days prior to enrollment (i.e., participant drug use must be stable prior to the study. They may not be enrolled if they began drug use within the past 60 days of assessment or if they intend to begin prescription drug use during the study); or
    * Systemic medication(s) (other than anti-histamines) that is known to cause ocular dryness (e.g. diuretics, anti-hypertensives, anti-depressants, hormone therapy) and whose dose of this medication(s) has not been stable within 30 days prior to enrollment. There must be no anticipated adjustments to the dose of these medications for the duration of the trial; or
    * Oral tetracyclines or azithromycin between enrollment and 30 days prior, unless their dosage will remain the same throughout the study; or
    * Topical ophthalmic antibiotics, anti-glaucoma medications, steroids, non-steroidal anti-inflammatory medications between enrollment and 30 days prior to enrollment, with the exception that patients who are newly prescribed short-term use (15 days or less) anti-inflammatories (e.g., corticosteroids) by the investigator during their screening visit may be included

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2023-03-07 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Mean change in basal tear secretion (Schirmer I test, with anesthesia) for designated study eye from baseline to Week 12 | 3 months
  Outcome reflects the volume of tears collected in the tear film over 5 minutes. A higher score reflects a larger tear film.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Amparo, MD, Principal Investigator — Independent
Locations (1):
- Córnea Atención Especializada, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No